CLINICAL TRIAL: NCT04824755
Title: A Prospective Study on Assessments of the Eye-related Quality of Life, Functional Vision, and Their Determinants Using the PedEyeQ in Children After Congenital Cataract Surgery and Their Families
Brief Title: Reduced ER-QOL in Families After Congenital Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yune Zhao (Other)
Responsible Party: Sponsor-Investigator, Yune Zhao, Director, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020080910
Record Dates: First submitted 2021-03-01; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Prospective Cross-sectional Study

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Demographics and clinic characteristics of children in different ages (Experimental)
  Interventions: Procedure: Yune Zhao
- PedEyeQ domain scores (Experimental)
  Interventions: Procedure: Yune Zhao
- Boxes represent first, median, and third quartile values. (Experimental)
  Interventions: Procedure: Yune Zhao
- Parent of kids aged 0-4y and 5-11y PedEyeQ domain scores (Experimental)
  Interventions: Procedure: Yune Zhao

INTERVENTIONS:
Procedure: Yune Zhao — Yune Zhao did congenital cataract surgeries

SUMMARY:
Children after congenital cataract surgery experience a lower quality of life and reduced functional vision. Their families have also been seriously affected. Investigators should pay more attention to them, and measures should be administered to families.

ELIGIBILITY:
Inclusion Criteria:

* visually not significant cataract, and ophthalmic surgery (incisional or laser) within one month

Exclusion Criteria:

* parents who were inability to communicate were also excluded

Ages: 0 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 166 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Gender of Child | through study completion, an average of half a year
  female,male
Parent/legal guardian Age | through study completion, an average of half a year
  under 25,26-30,31-35,36-40,over 41
Parent/legal guardian completing questionnaires | through study completion, an average of half a year
  father,mother,legal guardian
Native Place | through study completion, an average of half a year
  city,not the city
Parent/legal guardian highest level of education | through study completion, an average of half a year
  Primary school graduate,Junior-high graduate/technology secondary school graduate,high school graduate/junior college degree,College graduate,Postgraduate/professional degree
Staging operation | through study completion, an average of half a year
  primary IOL implantation, aphakia, secondary IOL implantation;using questionnaire and telephone follow-up
Postoperative timing | through study completion, an average of half a year
  Less than 1 year,1 to 2 years,2 to 3 years,More than 3 years;using questionnaire and telephone follow-up
Amblyopia treatment | through study completion, an average of half a year
  Cooperative,Average,Uncooperative,No treatment;using questionnaire and telephone follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmology and Optometry Hospital, Wenzhou, Zhejiang, China